CLINICAL TRIAL: NCT04843839
Title: Corneal Dystrophies Caused by SLC4A11 Mutation: A Promising New Paradigm Shift in Therapy Using an Ophthalmic Nonsteroidal Anti-Inflammatory Eye Drops
Brief Title: CHED - Congenital Hereditary Endothelial Dystrophy: New Paradigm Shift in Therapy Using Topical Eye Drops
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: L.V. Prasad Eye Institute (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, DR.MURALIDHAR, Consultant Pediatric Cornea and Anterior Segment services, LVPEI, L.V. Prasad Eye Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LEC-BHR-P-10-20-526
Record Dates: First submitted 2021-04-02; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Congenital Hereditary Endothelial Dystrophy of Cornea
Keywords: CHED
MeSH Terms: conditions — Corneal Dystrophy, Posterior Polymorphous, 1 | interventions — nepafenac; Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: Paired eye study- So one eye will be subjected to test drug, while the other eye will be subjected to a placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Eye (Experimental): These eyes will be given the Test drug, that is Nepafenac Eye Drops 0.1% w/v, at the dosage of 4 drops to be instilled in the eye 1 drop 4 times a day (every 4 hourly).That is at morning, afternoon, evening and at night. This is to be continued for a 6 months duration.
  Interventions: Drug: Nepafenac 0.1% Oph Susp
- Control Eye (Placebo Comparator): These eyes will be given the placebo, that is Carboxy-methylcellulose sodium lubricant eye drops 0.5%w/v, at the same dosage of 4 drops to be instilled in the eye 1 drop 4 times a day (every 4 hourly).That is at morning, afternoon, evening and at night. This is to be continued for a 6 months duration.
  Interventions: Drug: Refresh Tears 0.5% Lubricant Eye Drops

INTERVENTIONS:
Drug: Nepafenac 0.1% Oph Susp — Nepafenac 0.1% eye drops - Allergan : Dosage- 1 drop QID for 6 months
  Other Names: Amplinak
  Arms: Test Eye
Drug: Refresh Tears 0.5% Lubricant Eye Drops — Refresh Tears 0.5% w/v eye drops - Allergan : Dose- 1 drop QID for 6 months
  Other Names: Carboxy-methylcellulose sodium lubricant eye drops 0.5%w/v
  Arms: Control Eye

SUMMARY:
CHED- Congenital Endothelial Endothelial Dystrophy is a condition that causes corneal cloudiness.

Since, currently only surgery is being done to cure this condition, we are taking up the research of using topical eye drops for this condition which is a very simple and easy method.

Also, there are no significant side effects to this treatment.

DETAILED DESCRIPTION:
Introduction:

Corneal endothelial cell loss is often associated with blinding endothelial corneal dystrophies: relatively seen more frequently dominantly inherited (5%) FECD (Fuchs Endothelial Corneal Dystrophy) and rare recessive CHED1. Mutations of SLC4A11, an abundant corneal solute transporter, cause CHED and some cases of FECD. SLC4A11 is a unique member of the SLC4 family of bicarbonate transport proteins localized at the basolateral surface of corneal endothelial cells that contributes to osmotically-driven water flux from the stroma to aqueous humour to maintain corneal fluid-balance2.

While mutations and loss of functional SLC4A11 are reported to be associated with degeneration and death of endothelial cells, the detailed physiological roles of SLC4A11 still remain unknown. Seventy-eight different mutations, including 42- missense, 9- nonsense, 4- splice sites, and 23 insertion-deletion mutations, have been scattered across the gene reported in families with CHED from Indian populations3. Current therapeutic interventions Penetrating keratoplasty, Descemet's Stripping Automated Endothelial Keratoplasty (DSAEK), and Descemet's Membrane Endothelial Keratoplasty (DMEK) face problems such as shortage of donor corneas, complex surgical procedure, and incidence of graft failure in acute and chronic phases4, 5.

When studied in model cells, the most common molecular phenotype of mutant membrane proteins is mild misfolding. This biosynthetic defect renders the protein incapable of transit from the endoplasmic reticulum (ER) site of synthesis to its normal cellular location. Note that SLC4A11 localization in corneas of endothelial dystrophy patients has not been examined; the conclusion of ER retention presently rests on data from cell culture models. Correcting such biosynthetic defects is an attractive therapeutic approach for some genetic diseases affecting membrane proteins, best exemplified by the efficacy of the drug, Lumacaftor, in rescuing the cell-surface misfolded cystic fibrosis transmembrane conductance regulator (CFTR), the protein product of the cystic fibrosis (CF) gene.

Thus, there is an urgent need to find alternative therapy, which is reliable, simple and affordable. A lot of interest has being taken now a day in opting for a non-invasive way of modality over invasive ones. In SLC4A11 mutation corneal dystrophies, one such topic of interest is the hypothesized role of Non-Steroidal Anti-Inflammatory Drugs (NSAID's) as a medical management of corneal endothelial dystrophies.

Most SLC4A11 mutations lead to biosynthetic defects marked by accumulation of the protein in the Endoplasmic Reticulum, and their degradation before reaching the plasma membrane. This generated increased reactive oxygen species thus making the cell more vulnerable to oxidative and mitochondrial damage and more prone to apoptotic death.

A small-scale drug screen showed that Glafenine, a disused NSAID, was able to move some SLC4A11 mutants to the cell surface, suggesting that other NSAIDs might also have therapeutic potential.

Further, the retained protein in the Endoplasmic reticulum and the effects of various drugs on its expression to the surface was taken up by studies conducted by Alka et al on HEK293 cells expressing CHED and FECD mutation. They showed the efficacy of Diclofenac (Voltaren Ophthalmic) and Nepafenac over other NSAIDs in moving the endoplasmic reticulum-retained missense mutant SLC4A11 in 20 out of 30 test cells. Which showed a potential role of NSAIDs in these conditions.

This project is thus to screen NSAIDs available as eye drops for their ability to correct the cell-surfacing trafficking of SLC4A11 proteins.

Since their first introduction in ophthalmology, the use of NSAIDs have been exponentially expanded, from therapeutic applications including treatment of pain and inflammation associated with ophthalmic surgeries, to prevention and treat cystoid macular edema (CME) associated with cataract surgery, enhance mydriasis intraoperatively and in multiple inflammatory ophthalmic diseases, such as seasonal allergic conjunctivitis, viral conjunctivitis, uveitis, episcleritis and scleritis, as well as in retinal and choroidal diseases.

The main reason for this being that they are- (i) Easy to handle (ii) Non-invasive, (iii) Well-tolerated (iv) Sufficient ocular drug concentrations, while avoiding the systemic side effects associated with oral administration.

Nevertheless, the ocular drug bioavailability in the conventional topical formulations is notoriously poor, as only 1-5% of drug applied to the surface penetrates the cornea.

Besides these ocular anatomical and physiological constraints, another limiting factor encountered with anti-inflammatory drugs or immunosuppressive agents is their poor water solubility.

The prodrug approach is a chemical way to enhance drug permeability. The synthesized inactive prodrug exhibits a better corneal penetration and once in situ, is either chemically and/or enzymatically metabolized to become active. It was studied that, nepafenac, an amide prodrug of amfenac, belonging to the pharmacological NSAID class of aryl-acetic, in vitro demonstrated a nearly six-fold greater permeation coefficient than diclofenac.

In vivo, nepafenac easily crosses corneal and retinal tissues following topical ocular administration.

In this context, the study is intended in exploring the specific application of NSAID eye drops (Nepafenac) as a promising novel therapeutic approach for treating children with CHED.

There are no published reports of human trials for the application of NSAID eye drops in cases of Congenital Hereditary Endothelial Dystrophy.

Objectives:

To ascertain the clinical utility of topical ophthalmic NSAIDs in reversing or delaying the corneal cloudiness in children with CHED

Study Area/ Setting: Cornea and Anterior Segment Services, Kallam Anji Reddy campus, L V Prasad, Eye Institute, Hyderabad

Study Duration: 2 Years: 15th December 2020- 15th December 2022

Sample Size: Since it is a novel study with no other prior works, population size will be minimum 30 eyes

Study Population: Diagnosed cases of Congenital Hereditary Endothelial Dystrophy fulfilling the inclusion criteria

Study Design: Double-blinded, Placebo-controlled, Simple randomized control trial: A Paired eye study

Statistical Method: The data of this study will be compared by using the t-test or χ2 test depending if the data is parametric or non-parametric in nature

Methodology:

Targeting SLC4A11 mutation using ophthalmic NSAIDs preparation:

Test drug is Nepafenac eye drops 0.1%w/v. Given at the dosage of 4 drops to be instilled in the test eye 1 drop 4 times a day (every 4 hourly).That is at morning, afternoon, evening and at night. This is to be continued for a 6 months duration.

Control drug is Carboxy-methylcellulose sodium lubricant eye drops 0.5%w/v at the same dosage as the test eye drop but in the control eye.

The test eye will be chosen by Simple Randomization. For all the cases with an even serial number, the Right eye will be the test eye and for the odd numbered cases, the Left eye will be the test eye.

In order to ensure blinding of the patient and the investigators, both the drops will be dispensed in identical bottles and will be relabeled with the letter 'R' and 'L' signifying which eye the patient will be using them. This will be done in prior with only one member of the study having the list of the identity of drugs. The same person will also be providing the appropriately labeled drug for the patients and will not be a part of clinical evaluation and analysis of the patient's data.

To check for the patients' compliance, the patients will be required to get the used bottles at every visit and new ones will be provided. Since each bottle contains 5 ml of solution they would last for 25-30 days each, as will be our follow-up schedule for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Children upto 9 years of age diagnosed with CHED (Congenital Hereditary Endothelial Dystrophy) with bilaterally equal corneal involvement
* Patients agreeing on a regular monthly follow-up for a minimum of 6 months

Exclusion Criteria:

* Patient undergone any other surgery like Penetrating keratoplasty (PK), Descemet stripping automated endothelial keratoplasty (DSEK) and Descemet's membrane endothelial keratoplasty (DMEK), Glaucoma surgeries, in one of both eyes
* Patients with concomitant ophthalmic pathologies like glaucoma, poor corneal surface, dry eye disease, corneal ulcers, systemic inflammatory conditions, cataract, nystagmus, Reduced corneal sensation etc.
* Patients not able to come for follow-ups
* Asymmetrical corneal involvement
* Patients with known allergy to ophthalmic NSAID's
* Patients with asthma or bleeding dyscrasias
* Non-cooperative children

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Clinical change in the corneal transparency in the patients with CHED | Measured at each monthly follow-up till study completion, average 2 years
  Assessed by:
  Clinical grading of the corneal opacities at each visit as- Grade 0- no haze Grade 1-Iris details visible Grade 2-Pupil margin visible; iris details not visible Grade 3-Pupil margin not visible Grade 4-Cornea totally opaque
Change in the corneal transparency on Densitometry in the patients with CHED | Measured at each monthly follow-up till study completion, average 2 years
  Assessed by:
  Densitometry reading on Oculyzer machine

SECONDARY OUTCOMES:
Change in visual acuity in patients of CHED | Measured at each monthly follow-up till study completion, average 2 years
  Assessed by Subjective Refraction
Change in the Corneal thickness | Measured at each monthly follow-up till study completion, average 2 years
  Pachymetry/ Anterior Segment OCT (Optical Coherence Tomography) readings at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Muralidhar Ramappa, MS, Principal Investigator — L.V. Prasad Eye Institute; Neet Y Mehta, MBBS, Principal Investigator — L.V. Prasad Eye Institute
Locations (1):
- L V Prasad Eye Institute, Hyderabad, Banjara Hills, India